CLINICAL TRIAL: NCT04329052
Title: Promoting Mental Well-being for Secondary School Students Through an Experiential Learning Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UW18456
Record Dates: First submitted 2020-03-30; First posted 2020-04-01 (Actual); Last update posted 2020-04-01 (Actual); Status verified 2020-03

CONDITIONS: Mental Health
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Participants need to attend an adventure-based training with various experiential learning activities with a health educational talk on mental health.
  Interventions: Behavioral: Adventure-based training with health educational talk
- Control group (No Intervention): Participants would have their usual activity without any intervention.

INTERVENTIONS:
Behavioral: Adventure-based training with health educational talk — Participants need to attend an adventure-based training with various experiential learning activities with a health educational talk on mental health.
  Arms: Experimental group

SUMMARY:
Mental health problems in adolescents are a global problem and are becoming more prevalent in Hong Kong. Indeed, the rising incidence of emotional disturbances, adjustment and eating problems, depression, and suicidal tendencies have become major public health concerns.

Over the past few decades, Hong Kong has experienced a significant change in family structure, with an increase in small nuclear. Therefore, children may be overprotected by parents and become more fragile and less resilient to psychological distress, in the meantime, parents' high expectations for children's academic increase the pressure on the teenagers.

As resilience can promote better mental well-being with reduced anxiety and depressive symptoms, It is crucial for healthcare professionals to collaborate with youth centers in the community to build effective health promotion programs in schools that can enhance the resilience of adolescents and foster the development of their coping mechanisms and positive mental well-being so that adolescents can better combat mental health problems and lead healthier lives.

Adventure-based training rests on a theory of experiential learning, which involves a four-step model of concrete experience, reﬂective observation, abstract conceptualisation, and active experimentation. In adventure-based training, participants are required to join the activities which are psychologically and physically demanding. They may experience frustration and anxiety in the earlier stages, but this is potentially therapeutic as it can facilitate the process of concrete experience by encouraging them to accept an innovative approach in dealing with challenges. During the adventure process, the emphasis is placed on changing the dysfunctional and negative actions of team members into functional and positive actions, and on the interaction between team members in accomplishing different challenging tasks. Participants experience difficulties and look for possibilities, and with the proper guidance, facilitation and intervention of instructors the objectives of the training are achieved. Successful experience of this kind can facilitate the personal development and enhance the resilience and self-esteem of participants.

DETAILED DESCRIPTION:
Mental health problems in adolescents are a global problem and are becoming more prevalent in Hong Kong. Indeed, the rising incidence of emotional disturbances, adjustment and eating problems, depression, and suicidal tendencies have become major public health concerns.

Over the past few decades, Hong Kong has experienced a significant change in family structure, with small nuclear families gradually replacing extended families. Therefore, children receive more attention and may be overprotected by parents as a result of having fewer, if any, siblings. It is possible that this explains why children are more fragile, more vulnerable, and less resilient to psychological distress than were previous generations. Moreover, parents' high expectations for high academic achievement may also contribute to increased mental health problems among adolescents in Hong Kong. Most parents in Hong Kong believe that better careers and brighter futures are the inevitable results of higher academic achievement. Given this context, Hong Kong Chinese adolescents are exposed to considerable pressure within their families and schools while growing up.

Evidence suggests that depressive symptoms predict suicidal tendencies among children and adolescents. Although suicide rates in Hong Kong have dropped significantly from 18.8 per 100,000 in 2003 to 11.7 per 100,000 in 2016, a trend to increases in youth suicides in the past few years remains a concern. On the other hand, there is some evidence that resilience effectively prevents the development of mental health problems and is associated with positive mental health outcomes in adolescents, such as reduced levels of anxiety and depression [6]. It is therefore crucial for healthcare professionals to collaborate with youth centers in the community to build effective health promotion programs in schools that can enhance the resilience of adolescents and foster the development of their coping mechanisms and positive mental well-being so that adolescents can better combat mental health problems and lead healthier lives.

We conducted a 'proof-of-principle' randomised controlled trial on the effectiveness of experiential learning activity (adventure-based training programme) in promoting the psychological well-being of primary schoolchildren. This study provides some evidence that the adventure-based training programme is effective in enhancing self-esteem and reducing depressive symptoms among schoolchildren. Moreover, the study demonstrated the feasibility of implementing an adventure-based training programme in the Hong Kong Chinese context, with their content and nature shown to be acceptable to children and their parents.

Adventure-based training rests on a theory of experiential learning, which involves a four-step model of concrete experience, reﬂective observation, abstract conceptualisation, and active experimentation. It aims at changing cognitive thinking and behaviour, on different levels, through experience and practice in an outdoor environment. At the adventure-based training camp, participants would have a 'concrete experience' by having some physical activities. Trainers would observe and note down the important moments for further discussion and could recap the experiences that participants had had in the activity (reﬂective observation). While recapping the experience, trainers could assist the participants to sum up their experience and help them to discuss what they could do to make the experience better (abstract conceptualisation). With consolidation, the trainer would then encourage participants to think of similar situations that they might face in their daily lives and how they could apply the lessons learnt in this experience into others (active experimentation).

In adventure-based training, participants are required to join in different activities which are psychologically and physically demanding. They may experience frustration and anxiety in the earlier stages, but this is potentially therapeutic as it can facilitate the process of concrete experience by encouraging them to accept an innovative approach in dealing with challenges. During the adventure process, the emphasis is placed on changing the dysfunctional and negative actions of team members into functional and positive actions, and on the interaction between team members in accomplishing different challenging tasks. Participants experience difficulties and look for possibilities, and with the proper guidance, facilitation and intervention of instructors the objectives of the training are achieved. Successful experience of this kind can facilitate the personal development and enhance the resilience and self-esteem of participants.

ELIGIBILITY:
Inclusion Criteria:

* secondary school students from Form 1 to 3,
* able to speak Cantonese and read Chinese.

Exclusion Criteria:

* children with cognitive and learning problems identified from their school records.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 254 (Actual)
Dates: Start 2018-12-20 (Actual); Primary Completion 2019-11-25 (Actual); Study Completion 2019-11-25 (Actual)

PRIMARY OUTCOMES:
Change in resilience levels from baseline to 6-month follow-up between intervention and control group | 6-month follow-up
  The Resilience Scale-14 (RS-14) is a 14-item scale measuring personal competence, and acceptance of self and life. The item is answered using a 7-point Likert scale ranging from "strongly disagree" to "strongly agree," with total possible scores ranging from 14 to 98. Higher scores indicate higher levels of resilience.

SECONDARY OUTCOMES:
Resilience level at baseline | baseline
  The Resilience Scale-14 (RS-14) is a 14-item scale measuring personal competence, and acceptance of self and life. The item is answered using a 7-point Likert scale ranging from "strongly disagree" to "strongly agree," with total possible scores ranging from 14 to 98. Higher scores indicate higher levels of resilience.
Change in resilience levels from baseline to 1-month follow-up between intervention and control group | 1-month follow-up
  The Resilience Scale-14 (RS-14) is a 14-item scale measuring personal competence, and acceptance of self and life. The item is answered using a 7-point Likert scale ranging from "strongly disagree" to "strongly agree," with total possible scores ranging from 14 to 98. Higher scores indicate higher levels of resilience.
Depressive symptoms at baseline | baseline
  The Center for Epidemiologic Studies Depression Scale for Children (CES-DC) comprises 20 standardized items to evaluate depressive symptoms. All items are evaluated on a 4-point Likert scale in relation to their incidence during the previous week, and are scored from 0 to 3 (0 = not at all, 1 = a little, 2 = some, 3 = a lot); total possible scores thus range from 0 to 60, with higher scores indicating greater number of symptoms.
Change in depressive symptoms from baseline to 1-month follow-up between intervention and control group | 1-month follow-up
  The Center for Epidemiologic Studies Depression Scale for Children (CES-DC) comprises 20 standardized items to evaluate depressive symptoms. All items are evaluated on a 4-point Likert scale in relation to their incidence during the previous week, and are scored from 0 to 3 (0 = not at all, 1 = a little, 2 = some, 3 = a lot); total possible scores thus range from 0 to 60, with higher scores indicating greater number of symptoms.
Self-esteem levels at baseline | baseline
  The Rosenberg Self-esteem Scale (RSES) was designed to measure self-esteem as a global disposition and has been widely used with children [9]. The RSES consists of 10 items rated on a 4-point Likert scale ranging from 1 (strongly disagree) to 4 (strongly agree), with total possible scores ranging from 10 to 40. Higher scores indicate higher levels of self-esteem.
Change in self-esteem levels from baseline to 1-month follow-up between intervention and control group | 1-month follow-up
  The Rosenberg Self-esteem Scale (RSES) was designed to measure self-esteem as a global disposition and has been widely used with children [9]. The RSES consists of 10 items rated on a 4-point Likert scale ranging from 1 (strongly disagree) to 4 (strongly agree), with total possible scores ranging from 10 to 40. Higher scores indicate higher levels of self-esteem.
Change in depressive symptoms from baseline to 6-month follow-up between intervention and control group | 6-month follow-up
  The Center for Epidemiologic Studies Depression Scale for Children (CES-DC) comprises 20 standardized items to evaluate depressive symptoms. All items are evaluated on a 4-point Likert scale in relation to their incidence during the previous week, and are scored from 0 to 3 (0 = not at all, 1 = a little, 2 = some, 3 = a lot); total possible scores thus range from 0 to 60, with higher scores indicating greater number of symptoms.
Change in self-esteem levels from baseline to 6-month follow-up between intervention and control group | 6-month follow-up
  The Rosenberg Self-esteem Scale (RSES) was designed to measure self-esteem as a global disposition and has been widely used with children [9]. The RSES consists of 10 items rated on a 4-point Likert scale ranging from 1 (strongly disagree) to 4 (strongly agree), with total possible scores ranging from 10 to 40. Higher scores indicate higher levels of self-esteem.

CONTACTS AND LOCATIONS:
Overall Officials: Ho Cheung William Li, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No